CLINICAL TRIAL: NCT04018378
Title: An Open-label, Randomized, Single-dose Crossover Study to Evaluate the Pharmacokinetics, Safety and Tolerability of HIP1502 in Healthy Male Subjects
Brief Title: A Clinical Study to Evaluate the Pharmacokinetics, Safety and Tolerability of HIP1502
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Ji-Young Park, Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-VANC-101
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Healthy
MeSH Terms: interventions — Varenicline

STUDY DESIGN:
Intervention Model Description: an open-label, randomized, single-dose crossover clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RT (Experimental): period 1: HGP1604 1mg (reference drug, R) will be administered once orally.
  period 2: HIP1502 1mg (test drug, T) will be administered once orally after 14 days of the washout period.
  Interventions: Drug: varenicline tartrate 1mg (HGP1604, R) - varenicline oxalate 1mg (HIP1502, T), RT
- TR (Experimental): period 1: HIP1502 1mg (test drug, T) will be administered once orally.
  period 2: HGP1604 1mg (reference drug, R) will be administered once orally after 14 days of the washout period.
  Interventions: Drug: varenicline oxalate 1mg (HIP1502, T) - varenicline tartrate 1mg (HGP1604, R), TR

INTERVENTIONS:
Drug: varenicline tartrate 1mg (HGP1604, R) - varenicline oxalate 1mg (HIP1502, T), RT — varenicline tartrate 1mg (HGP1604) was used as a reference drug and varenicline oxalate 1mg (HIP1502) was used as a test drug.
  Arms: RT
Drug: varenicline oxalate 1mg (HIP1502, T) - varenicline tartrate 1mg (HGP1604, R), TR — varenicline tartrate 1mg (HGP1604) was used as a reference drug and varenicline oxalate 1mg (HIP1502) was used as a test drug.
  Arms: TR

SUMMARY:
The clinical trial aims to assess the pharmacokinetics, safety and tolerability of HIP1502 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers aged between ≥20 and ≤45 years old
2. Weight ≥ 50 kg, with calculated body mass index (BMI) of ≥ 18 and ≤ 29.9 kg/m2
3. Subject who voluntarily agrees to participate in this study and signs the informed consent form.

Exclusion Criteria:

1. History or presence of clinically significant and active cardiovascular, respiratory, hepatobiliary, renal, hematological, oncological, urinary, psychiatric, gastrointestinal, endocrine, immune, dermatologic or neurologic disorder.
2. With symptoms indicating acute illness within 28 days prior to the first IP administration.
3. Any medical history that may affect drug absorption, distribution, metabolism, and excretion.
4. Any clinically significant activity of chronic medical illness.
5. History of any clinically significant allergic reaction including induced by varenicline (However, mild allergic rhinitis or allergic dermatitis which do not require medication could be included).
6. Positive blood tests for HBs Ag, anti-HCV Ab, anti-HIV Ab, or VDRL.
7. Use of any prescription drugs and herbal preparations within 14 days prior to study drug administration or use of over-the-counter medications (OTC) and vitamin products within 10 days prior to study drug administration.
8. Inability to take standard hospital diet.
9. Donation of blood within 60 days prior to study drug administration or apheresis within 20 days, or blood transfusion within 30 days prior to the first IP administration.
10. Exposure to any investigational drug or placebo within 90 days prior to the last IP administration.
11. Subjects with excessive caffeine intake (more than 5 cups/day), heavy or regular alcohol intake (more than 210 g/week).
12. Any use of tobacco or nicotine within three months.
13. Subjects rejected to use clinically effective contraceptive methods during the study period.
14. Subjects having been deemed inappropriate for the trial as determined by the investigator.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2018-09-17 (Actual)

PRIMARY OUTCOMES:
AUC | 0 (predose) ~ 96 hours
  area under the plasma concentration-time curve
Cmax | 0 (predose) ~ 96 hours
  maximum plasma concentration of the drug

SECONDARY OUTCOMES:
Tmax | 0 (predose) ~ 96 hours
  time to maximum plasma concentration
T1/2 | 0 (predose) ~ 96 hours
  terminal elimination half-life
CL/F | 0 (predose) ~ 96 hours
  apparent total body clearance of the drug from plasma
Vd/F | 0 (predose) ~ 96 hours
  apparent volume of distribution

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Clinical Pharmacology & Toxicology, Anam Hospital, Korea University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No